CLINICAL TRIAL: NCT03835351
Title: Urinary Retention After Laparoscopic Inguinal Hernia Repair: A Randomized Controlled Trial Comparing Intraoperative Urinary Catheter Versus no Catheter
Brief Title: Urinary Retention After Laparoscopic Inguinal Hernia Repair: Comparing the Use of the Intraoperative Urinary Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Michael Rosen, Director of the Comprehensive Hernia Center, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-070
Record Dates: First submitted 2019-02-07; First posted 2019-02-08 (Actual); Results first posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Inguinal Hernia
Keywords: Urinary catheter; Urinary retention; Laparoscopic inguinal hernia repair
MeSH Terms: conditions — Hernia, Inguinal; Urinary Retention | interventions — Urinary Catheters; Urinary Catheterization

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intraoperative urinary catheter (Other): After induction of general anesthesia, a standard catheterization kit available at the institution where the surgery is being performed will be used to place the urinary catheter using standard sterile technique.
  Interventions: Device: Urinary Catheter
- No intraoperative urinary catheter (No Intervention): No intraoperative urinary catheter will be used during the case

INTERVENTIONS:
Device: Urinary Catheter — An intraoperative urinary catheter will be inserted which will be taken out at the end of the case
  Other Names: Foley
  Arms: Intraoperative urinary catheter

SUMMARY:
This will be a randomized controlled study which will compare the rate of post-operative urinary retention after laparoscopic inguinal hernia repair between patients who receive an intra-operative urinary catheter and those who do not. The primary aim of the study is to determine if the use of intra-operative urinary catheter reduces the incidence of post-operative urinary retention after laparoscopic inguinal hernia repair. Specific patient inclusion criteria include all patients aged 18 years or older presenting for an elective unilateral or bilateral inguinal hernia repair, who are able to tolerate general anesthesia and are considered eligible to have a hernia repair through a laparoscopic approach.

DETAILED DESCRIPTION:
An inguinal hernia repair is a common outpatient procedure with a low rate of morbidity. One well-recognized complication of this operation is post-operative urinary retention (PUR), which is a failure of spontaneous voiding requiring insertion of a urinary catheter. The reported incidence of PUR ranges between 0.4 and 3% of open tension-free repairs. For laparoscopic inguinal hernia repairs that range is between 1 and 22. Since no randomized controlled trials have evaluated PUR as the primary outcome exist in literature, there is no consensus on whether catheter use aids in minimizing post-operative urinary retention. Routine use of intraoperative catheterization increases the risk of urethral trauma, catheter-associated infections and bladder damage leading to increased cost of care and potential patient morbidity. On the other hand, PUR is associated with additional procedures, such as catheterization, which may delay hospital discharge or increase the length of stay and cause patient discomfort. This work aims to study the effect of intraoperative catheters on PUR and whether the aforementioned risks associated with this procedure are justified.

We hypothesize that the use of intra-operative urinary catheter reduces the incidence of postoperative urinary retention after laparoscopic inguinal hernia repair, thus justifying the potential complications associated with intra-operative catheter insertion.

All patients will be asked to void in the pre-operative area prior to going into the operating room. Patients will be operated in the supine, and slight Trendelenburg position (15º degrees), with arms tucked along the body. The procedure will be performed under general anesthesia. After induction of anesthesia, randomization will occur. It will be performed according to a computer-generated block randomization scheme. The randomization will be stratified for unilateral or bilateral hernias. Antibiotic prophylaxis will be performed according to institutional protocol. Pharmacological prophylaxis of venous thromboembolic events is usually not necessary for general laparoscopic inguinal hernia repair. Although, if deemed necessary, this will be performed per Surgical Care Improvement Project (SCIP) protocol and will not be considered a protocol deviation. Skin preparation and hair removal will be performed per SCIP protocol. All necessary materials, including the urine catheterization kit, will be available in the operative room before the start of the procedure.

The Americas Hernia Society Quality Collaborative (AHSQC) registry will serve as the main platform for data collection. Registry-based trials use data available in a preexisting database to increase the efficiency of performing RCTs, decreasing the high cost and logistical challenges associated with operationalizing this type of research. Post-operative urinary retention will be defined as post-operative failure to void requiring straight catheterization, placement of an indwelling catheter or return to the emergency department due to failure to void after discharge from the hospital. Bladder scanning, its timing and specific criteria for placement of urinary catheter will be determined by the standard policies of each institution where the surgery was performed and the surgeon.

Specific Aim #1: To determine if the use of intra-operative urinary catheter reduces the incidence of postoperative urinary retention after laparoscopic inguinal hernia repair. This will be assessed by comparing the PUR rates between the two study groups.

Specific Aim #2: To determine if there is a difference in the rates of intraoperative bladder injuries between the study groups. This will be determined by comparing the rates of intraoperative bladder injuries between the two study groups.

Specific Aim #3: To determine the rate of urinary tract complications after insertion of the intra operative urinary catheter for the control group. This will be accomplished by analyzing the rates of urinary tract injury, infections and bladder injuries due to intraoperative catheter placement.

Specific Aim #4: To determine the rate of urinary tract complications after insertion of a urinary catheter for patients who develop PUR. This will be accomplished by analyzing the rates of urinary tract injury, or infections and bladder injuries due to catheter placement after patients develop PUR.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent
* Unilateral or bilateral inguinal hernia
* Scheduled for elective inguinal hernia repair
* Eligible to tolerate general anesthesia
* Eligible to undergo minimally invasive inguinal hernia repair

Exclusion Criteria:

* Diagnosed with benign prostate hyperplasia (BPH)
* Younger than 18 years old
* Unable to give informed consent
* Emergent inguinal hernia repairs ( acute incarceration or strangulation)
* Unable to tolerate general anesthesia
* Not eligible for minimally invasive inguinal hernia repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rosen, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Comprehensive Hernia Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, rather the results of the aggregate groups of patients will be shared

REFERENCES:
- [Background] Koch CA, Grinberg GG, Farley DR. Incidence and risk factors for urinary retention after endoscopic hernia repair. Am J Surg. 2006 Mar;191(3):381-5. doi: 10.1016/j.amjsurg.2005.10.042. PMID 16490551
- [Background] Jensen P, Mikkelsen T, Kehlet H. Postherniorrhaphy urinary retention--effect of local, regional, and general anesthesia: a review. Reg Anesth Pain Med. 2002 Nov-Dec;27(6):612-7. doi: 10.1053/rapm.2002.37122. PMID 12430114
- [Background] Blair AB, Dwarakanath A, Mehta A, Liang H, Hui X, Wyman C, Ouanes JPP, Nguyen HT. Postoperative urinary retention after inguinal hernia repair: a single institution experience. Hernia. 2017 Dec;21(6):895-900. doi: 10.1007/s10029-017-1661-4. Epub 2017 Sep 4. PMID 28871414
- [Background] Patel JA, Kaufman AS, Howard RS, Rodriguez CJ, Jessie EM. Risk factors for urinary retention after laparoscopic inguinal hernia repairs. Surg Endosc. 2015 Nov;29(11):3140-5. doi: 10.1007/s00464-014-4039-z. Epub 2015 Jan 1. PMID 25552230
- [Background] Sivasankaran MV, Pham T, Divino CM. Incidence and risk factors for urinary retention following laparoscopic inguinal hernia repair. Am J Surg. 2014 Feb;207(2):288-92. doi: 10.1016/j.amjsurg.2013.06.005. Epub 2013 Nov 5. PMID 24200291
- [Background] Muysoms FE, Vanlander A, Ceulemans R, Kyle-Leinhase I, Michiels M, Jacobs I, Pletinckx P, Berrevoet F. A prospective, multicenter, observational study on quality of life after laparoscopic inguinal hernia repair with ProGrip laparoscopic, self-fixating mesh according to the European Registry for Abdominal Wall Hernias Quality of Life Instrument. Surgery. 2016 Nov;160(5):1344-1357. doi: 10.1016/j.surg.2016.04.026. Epub 2016 Jun 14. PMID 27316825
- [Background] Arnold MR, Coakley KM, Fromke EJ, Groene SA, Prasad T, Colavita PD, Augenstein VA, Kercher KW, Heniford BT. Long-term assessment of surgical and quality-of-life outcomes between lightweight and standard (heavyweight) three-dimensional contoured mesh in laparoscopic inguinal hernia repair. Surgery. 2019 Apr;165(4):820-824. doi: 10.1016/j.surg.2018.10.016. Epub 2018 Nov 16. PMID 30449696
- [Derived] Woo KP, Ellis RC, Maskal SM, Remulla D, Shukla P, Rosen AJ, Wetzka I, Osei-Koomson W, Phillips S, Miller BT, Beffa LR, Petro CC, Krpata DM, Prabhu AS, Menzo EL, Rosen MJ. The association of permanent versus absorbable fixation on developing chronic post-herniorrhaphy groin pain in patients undergoing laparoscopic inguinal hernia repair. Surg Endosc. 2024 Jun;38(6):3433-3440. doi: 10.1007/s00464-024-10866-z. Epub 2024 May 6. PMID 38710888
- [Derived] Fafaj A, Lo Menzo E, Alaedeen D, Petro CC, Rosenblatt S, Szomstein S, Massier C, Prabhu AS, Krpata DM, Cha W, Montelione K, Tastaldi L, Alkhatib H, Zolin SJ, Okida LF, Rosen MJ. Effect of Intraoperative Urinary Catheter Use on Postoperative Urinary Retention After Laparoscopic Inguinal Hernia Repair: A Randomized Clinical Trial. JAMA Surg. 2022 Aug 1;157(8):667-674. doi: 10.1001/jamasurg.2022.2205. PMID 35704302

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intraoperative Urinary Catheter | No Intraoperative Urinary Catheter
Started | 241 | 250
Completed | 241 | 250
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intraoperative Urinary Catheter | No Intraoperative Urinary Catheter | Total
Number analyzed (Participants) | 241 | 250 | 491
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 61 [52 to 68] | 62 [49 to 69] | 61 [51 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 17 | 26
  Male | 232 | 233 | 465
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Pacific Islander | 4 | 3 | 7
  Black, not of Hispanic Origin | 18 | 33 | 51
  Hispanic | 5 | 9 | 14
  Middle Eastern | 5 | 1 | 6
  White, not of Hispanic Origin | 209 | 204 | 413
Region of Enrollment [Number; unit: participants]
  United States | 241 | 250 | 491

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Post Operative Urinary Retention
Description: The rate of postoperative urinary retention requiring insertion of a urinary catheter
Time Frame: From the day of surgery until postoperative day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Intraoperative Urinary Catheter | No Intraoperative Urinary Catheter
Number analyzed (Participants) | 241 | 250
Participants | 23 | 21

2. Secondary Outcome: Number of Participants With Intraoperative Bladder Injuries
Description: This will be determined by comparing the rates of intraoperative bladder injuries between the two study groups
Time Frame: Measured from Beginning of Anesthesia to the End of Anesthesia and up to 4 hours Post Operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Intraoperative Urinary Catheter | No Intraoperative Urinary Catheter
Number analyzed (Participants) | 241 | 250
Participants | 0 | 0

3. Secondary Outcome: Number of Participants Who Have Complications From Intra-operative Urinary Catheter
Description: This will be accomplished by analyzing the rates of urinary tract injury, infections and bladder injuries due to intraoperative catheter placement.
Time Frame: From the day of surgery until postoperative day 30
Measure: Number; unit: participants
Arm/Group | Intraoperative Urinary Catheter | No Intraoperative Urinary Catheter
Number analyzed (Participants) | 241 | 250
participants
  Intraop Complication Urethral Trauma | 1 | 0
  Intraop Complication, other | 5 | 1

4. Secondary Outcome: Number of Participants With Complications Urinary Catheter Who Develop Retention
Description: This will be accomplished by analyzing the rates of urinary tract injury, or infections and bladder injuries due to catheter placement after patients develop post operative urinary retention.
Time Frame: From the day of surgery until postoperative day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Intraoperative Urinary Catheter | No Intraoperative Urinary Catheter
Number analyzed (Participants) | 241 | 250
Participants
  Urinary Tract Injury | 1 | 0
  Bladder Injuries | 0 | 0
  Infection | 21 | 28
  None | 219 | 222

ADVERSE EVENTS:
Time Frame: 30 days following surgery
Arm/Group | Intraoperative Urinary Catheter | No Intraoperative Urinary Catheter
All-Cause Mortality (participants affected / at risk) | 0/241 | 0/250
Serious Adverse Events (participants affected / at risk) | 1/241 | 0/250
Other Adverse Events (participants affected / at risk) | 3/241 | 11/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intraoperative Urinary Catheter (N=241) | No Intraoperative Urinary Catheter (N=250)
Urethra Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intraoperative Urinary Catheter (N=241) | No Intraoperative Urinary Catheter (N=250)
Anemia Requiring Transfusion (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT03835351/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT03835351/ICF_001.pdf